CLINICAL TRIAL: NCT03085355
Title: Evaluation of the Effects of the Association of the Osteopathic Manipulative Treatment to Exercises, Education for Pain in Participants With Cervical Pain - Pragmatic Clinical Trial Randomized
Brief Title: Evaluation of the Effect of the OMT Exercises Education for Pain in Participants With Cervical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Osteopatia (Other)
Responsible Party: Principal Investigator, Sandro Groisman, PT, DO, MSc, Master, Instituto Brasileiro de Osteopatia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Neck Pain; Pain, Neck
Keywords: neck pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise; Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises and PNE (Active Comparator): Individuals with neck pain will receive a exercises program and pain neuroscience education. Participants will receive treatments during 4 weeks, 1 treatment per week
  Interventions: Procedure: Exercises and PNE
- Osteopathic manipulative treatment (Experimental): Individuals with neck pain in this group will also receive a exercises program and pain neuroscience education and the participants will receive treatments during 4 weeks, 1 treatment per week associated with Osteopathic Manipulative Treatment (OMT)
  Interventions: Procedure: Osteopathic manipulative treatment

INTERVENTIONS:
Procedure: Exercises and PNE — Exercise for stretching and strength for neck muscles and pain neuroscience education
  Arms: Exercises and PNE
Procedure: Osteopathic manipulative treatment — Osteopathic manipulative treatment associated exercise for stretching and strength for neck muscles and pain neuroscience education
  Arms: Osteopathic manipulative treatment

SUMMARY:
The purpose of this randomized pragmatic clinical trial is to assess the effectiveness of the association of the osteopathic manipulative treatment in individuals with chronic non-specific neck pain who receive a exercice program and pain neurocience education.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether osteopathic manipulative treatment associated exercises and pain neurocience education improves pain and function in individuals with chronic non-specific neck pain

Design: a randomized single blind controlled pragmatic trial will be conducted trial. Patients (n=40) with non-specific neck pain will be randomized to receive 1) osteopathic manipulative treatment and exercise and and pain neurocience education (n=20) or 2) exercise alone and pain neurocience education (n=20). Participants will receive 8 treatments during 4 weeks. Clinical outcomes will be obtained at 1 week, four weeks and 24 weeks after end of treatment.

Methods:

The primary outcome will be pain measured by 11-point numerical pain rating scale. The secondary outcome will be disability measured by the Neck Disability Index, range of motion measured by Cervical Range of Motion device, Pressure pain threshold measured by electronic algometer, global perceived effect, Pain Self-Efficacy Questionnaire and pain catastrophizing scale

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of chronic neck pain does not specify that persists for more than 3 months
* Pain at least 3 points on 0-10 numeric pain rating and at least 14% disability on Neck Disability Index

Exclusion Criteria:

* individuals who report inflammatory previous surgery, spondylolisthesis, spinal stenosis, herniated disc, radiculopathy, fracture and musculoskeletal degenerative diseases. , Cancer, neurological diseases, pregnancy. They will be excluded participants who received some form of manipulative treatment in the last three months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measured by numeric rating scale

SECONDARY OUTCOMES:
Functionality and disability | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measured by Neck Disability Scale
Range of motion | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measured by CROM device
Pressure pain threshold | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measured by electronic algometer
Global perceived effect | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measured by global perceived rating scale
Self-efficacy | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measured by The Pain Self-Efficacy Questionnaire
Catastrophizing | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measure by pain catastrophizing scale
kinesiophobia | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measure by TAMPA scale
McGuill | Measured pre and post treatment, 4 weeks after treatment and 8 weeks after treatment
  measure by Mcguill scale

CONTACTS AND LOCATIONS:
Overall Officials: sandro Groisman, Principal Investigator — UFCSPA Federal University of Health Science of Porto Alegre; Geraldo Jotz, Phd, Study Director — UFCSPA Federal University of Health Science of Porto Alegre
Locations (1):
- Sandro Groisman, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No